CLINICAL TRIAL: NCT00221949
Title: Development of a Comprehensive Study of the Peripheral Nerves in the Lower Arm and Lower Leg Using an Ultrasound Guided Approach
Brief Title: Visualizing Peripheral Nerves Using Ultrasound-Guided Approach
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: UHN05-0491-AE
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2005-08

CONDITIONS: Regional Anesthesia
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Ultrasound

SUMMARY:
Peripheral nerve blocks of the limbs are very useful in providing anesthesia and pain relief for orthopedic procedures in the limbs (elbows, arms, knees, and legs). Considering that current nerve block techniques involve locating the main nerves at the top of the limb and "freezing" those neural structures in order to provide pain relief to the rest of the extremity, a comprehensive study of the nerves located lower in the limbs is needed. This study provides a step in the direction of the development of techniques for advanced nerve blockade that target nerve structures lower in the limbs to provide precise pain relief rather than widespread numbness.

The objective of the study aims to use direct ultrasound guidance to develop a comprehensive examination and identification of the peripheral nerves in the lower region of the upper and lower limbs (arms and legs). In a sense, this process allows us to "visualize" the nerves. In the future, with the experience of visualizing these nerves with the ultrasound machine, we can develop techniques that may allow us to perform anesthetic blockade with greater success and fewer complications.

An ultrasound exam will be performed on 8 healthy volunteers to view the peripheral nerves in the lower arm in three locations: the elbow area, the wrist area, and the midpoint of the arm between the elbow and the wrist. A set of 8 healthy patients will be given an ultrasound exam to view the peripheral nerves located in the lower leg by imaging three locations: the knee area, the ankle area, and the midpoint of the leg between the knee and the ankle. The appropriate nerves will be identified by ultrasound and images will be captured and recorded for further corroboration. The group of 16 subjects will allow for varied observations of anatomical positions of neural and vascular structures, while keeping the sample size fairly small. No injections will be made at any time during this study.

DETAILED DESCRIPTION:
The nerves of the upper extremities derive from the brachial plexus, and likewise, the nerves of the lower extremities derive from the lumbo-sacral plexus (1). In clinical practice, nerve blocks are commonly performed to provide postoperative analgesia after orthopedic procedures involving the upper and lower extremities (2,3). They may also be used as a sole anesthetic technique during surgery.

The two main concerns with upper and lower extremity blocks, as with other regional anesthetic techniques, are technical failure and block related complications. The most cited complications are bleeding from inadvertent arterial or venous puncture, intravascular injection of local anesthetic resulting in central nervous system or cardiac toxicity, and intraneural injection of local anesthetic resulting in peripheral neuropathy of varying degrees (4,5).

Both technical failures and complications are related at least in part, to the fact that all the techniques used to date are blind. Anatomical landmarks (as described in the literature) and nerve stimulators are helpful ways to localize the nerves to be blocked.

We believe that the best approach to improve success rate and minimize complications of peripheral nerve blocks is to use image-guided techniques. In the last few years, different imaging modalities have been used to evaluate the peripheral nerves of the upper and lower extremities. Studies currently underway at our institution seek to develop a comprehensive technique for upper and lower extremity nerve blocks. However, this involves anesthetizing from the top of the limb in order to numb the entire extremity. More research is needed to derive a comprehensive examination of the peripheral nerves found in the lower regions of the upper and lower extremities. While CT scanning and MRI are probably the techniques of choice when it comes to diagnosing nerve pathology, they would not be useful in the perioperative setting due to the lack of portability and the inability to perform real time imaging simultaneously with nerve block performance (6,7).

Ultrasound has been used successfully in the last few years to image the peripheral nerves of the upper extremity (8,9). The development of higher frequency ultrasound probes, and higher imaging resolution has made it possible to localize and evaluate peripheral nerves with ultrasound, something that was not possible only 10-15 years ago. The anatomy of the brachial plexus has been described by a number of authors. There have been some preliminary studies looking into the possibility of developing a real-time ultrasound guided technique for upper extremity blocks (10, 11, 12, 13,). Studies performed at our institution involving refining a technique for upper extremity blocks show encouraging results.

It is clear, that ultrasound can be used to a further degree of sophistication in order to image peripheral nerves in the lower parts of the upper and lower limbs. As expressed by many of the referenced authors, ultrasound use is likely to increase significantly in the coming years, both in the areas of diagnostic radiology and clinical regional anesthesia, to guide nerve blocks (17). As a result, it is evident that the development of an advanced technique for anesthetic blockade - which targets a precise location or nerve - can derive from this knowledge and recognition of peripheral nerves located in the lower parts of limbs. To this date, nonetheless, there is no systematic evaluation of the nerves located in the lower regions of the upper and lower limbs by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* 16 health volunteers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada